CLINICAL TRIAL: NCT03540979
Title: Endometrial Preparation With Aromatase Inhibitors Versus Estradiol in Frozen Embryo Transfer Cycles
Brief Title: Endometrial Preparation in Frozen Embryo Transfer Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC180016-18CTIL
Record Dates: First submitted 2018-02-08; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Reproductive Behavior
MeSH Terms: conditions — Reproductive Behavior | interventions — Letrozole; Ovidrel; estradiol, estriol drug combination; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estrogen (Active Comparator): Endometrial preparation: Estrogen supplements (Estradiol 6mg/d) will be started at the 2nd-3rd day of the cycle. First US scan will be performed after 10 days. If necessary, adjusting the estradiol doses will be performed according to the physician decision. After achieving trilinear endometrial thickness ≥8mm progesterone supplements (Endometrin 100mg*3/d) will be administrated. Embryo transfer will be performed after completing 5 days of progesterone supplements (at the 6th day after starting the progesterone supplements).
  Interventions: Procedure: endometrial preparation for frozen blastocyst transfer; Drug: Estrofem; Drug: Endometrin 100Mg Vaginal Insert
- Letrozole (Experimental): Women in the Letrozole arm will be treated with Aromatase inhibitors ( Letrozole; 2.5 mg per day) starting at the 3rd day of the cycle for 5 days. US scan,and blood work for serum Estradiol (E2) and progesterone (P) will initially be examined 3-5 days after the last Letrozole pill. Following US scans and serum E2+P will be performed according to the treating physician decision. When US scan demonstrate trilaminar endometrium ≥8 mm and the dominant follicle will be ≥18mm, hCG will be administrated ( recommbinant hCG - Ovitrelle 250 mcg) and 3 days later vaginal Endometrin 100mg*3/d will be started. Single vitrified-warmed blastocyst transfer will be performed after completing 4 days of the progesterone supplements (7 days from hCG administration).
  Interventions: Procedure: endometrial preparation for frozen blastocyst transfer; Drug: Letrozole; Drug: Ovidrel; Drug: Endometrin 100Mg Vaginal Insert

INTERVENTIONS:
Procedure: endometrial preparation for frozen blastocyst transfer — medical endometrial preparation for frozen blastocyte transfer
Drug: Letrozole — Aromatase inhibitor - 2.5mg/d for 5 days
  Other Names: Femara
  Arms: Letrozole
Drug: Ovidrel — recommbinant hCG 250 mcg- single sc injection to induce ovulation
  Other Names: Ovidre
  Arms: Letrozole
Drug: Estrofem — Estrofem 2mg*3/d for endometrial preparation
  Other Names: Estrsdiol
  Arms: Estrogen
Drug: Endometrin 100Mg Vaginal Insert — vaginal tab for lutheal support

SUMMARY:
Comparison of protocols for frozen embryo transfer (ET): One protocol using Estrogen supplements and the second protocol using Letrozole

DETAILED DESCRIPTION:
Study design. Randomized control trial will be conducted at the IVF Units at Meir Medical Center.

Participants. Patients undergoing frozen embryo transfer (ET) cycle with single blastocyst transfer.

Outcome measures The primary outcome measure is clinical pregnancy rate defined as intrauterine pregnancy with positive fetal heart beat measured 2-3 weeks after positive β-hCG test. Secondary outcome measures include: pregnancy rate (defined as positive beta-hCG test 12-14 days after embryo transfer), implantation rate and miscarriage rate.

Methods.

Patients who are candidates for vitrified-warmed single blastocyst transfer will be recruited for the study after signing informed consent form. Patients will then be randomized to one of the following groups:

The Letrozole group (study group); Women in the Letrozole arm will be treated with Aromatase inhibitors (Letrozole; 2.5 mg per day) starting on the 3rd day of the cycle for 5 days. US scan, blood work for serum Estradiol (E2) and progesterone (P) will initially be examined 3-5 days after the last Letrozole pill. Additional US scans and serum E2+P will be performed according to the treating physician's decision. When US scan demonstrates trilaminar endometrium ≥8 mm and the dominant follicle will be ≥18mm, Human Chorionic Gonadotropin (hCG) will be administred(recommbinant hCG - Ovitrelle 250 mcg) and 3 days later vaginal Endometrin 100mg*3/d will be started. Single vitrified-warmed blastocyst transfer will be performed after completing 4 days of the progesterone supplements (7 days from hCG administration). Patients will continue with progesterone supplements untill a pregnancy test which will be performed 12 days following the embryo transfer. If the pregnancy test comes out positive another test will be administered 2 days later, and viability US scan will be performed 2 weeks later. Luteal support will be taken untill the 9th week of pregnancy.

The Estrogen-Progesterone group (control group):

Endometrial preparation: Estrogen supplements (Estradiol 6mg/d) will start at the 2nd-3rd day of the cycle. First US scan will be performed after 10 days. If necessary, adjusting the estradiol doses will be performed according to the physician's decision. After achieving trilinear endometrial thickness ≥8mm progesterone supplements (Endometrin 100mg*3/d) will be administrated. Embryo transfer will be performed after completing 5 days of progesterone supplements (at the 6th day after starting the progesterone supplements). Patients will continue with progesterone supplements untill pregnancy test which will be performed 12 days following the embryo transfer. If pregnancy test is positive another test will be performed 2 days later, and viability US scan will be performed 2 weeks later. Luteal support will be taken untill the 9th week of pregnancy.

Sample size estimation In order to obtain a significance of 0.05 and a power of 80%, the investigators require 54 patients per group (total 108). This estimation is based on the live birth rate of 30% at the estrogen-progesterone endometrial preparation group compared to 60% at the letrozole preparation group. However, the investigators plan to recruit 100 patients in each group due to cycles with lost to follow up and ET cancellation.

Statistical Analysis:

The investigators will use the Shapiro Wilks test to evaluate the distribution of the data. Comparisons will be analyzed using Student's T test or Mann-Whitney U test when appropriate. Proportions will be compared with Chi Square test or Fisher exact test. P value of less than 0.05 will be considered significant. Multivariate logistic regression analysis will be used to compare continuous variables, while controlling for multiplicity and confounding factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing frozen embryo transfer cycle
2. Single blastocyst transfer
3. Normal uterine cavity.

Exclusion criteria:

1. Woman age older than 40
2. Cleavage stage embryo
3. More than 3 previous transfers w/o pregnancy
4. Oocyte donation cycle.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy | 4 to 5 weeks after the embryo transfer ( 6-7 weeks of pregnancy).
  The primary outcome measure is clinical pregnancy rate defines as intrauterine pregnancy with positive fetal heart beat measure 2-3 weeks after positive β-hCG TEST ( 6-7 weeks of pregnancy)

SECONDARY OUTCOMES:
pregnancy rate | 12-14 days after the embryo transfer
  Secondary outcome measures include: pregnancy rate (defines as positive beta-hCG test 12-14 days after embryo transfer),

IPD SHARING:
Plan to Share IPD: No